CLINICAL TRIAL: NCT07228000
Title: Bundled Cancer Screening and Genetic Services Navigation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 24-08-699; R01CA301168 (NIH)
Record Dates: First submitted 2025-11-12; First posted 2025-11-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Screening; Colon Cancer Screening; Genetics Predisposition
Keywords: navigation; mammography; colonoscopy; Fecal Immunochemical Test; genetic testing; risk assessment
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Usual care breast cancer screening navigation (Experimental)
  Interventions: Behavioral: Breast cancer screening navigation
- Multicancer screening navigation (Experimental)
  Interventions: Behavioral: Multicancer screening navigation
- Usual care breast cancer screening navigation + usual care genetic referral (Experimental)
  Interventions: Behavioral: Breast cancer screening navigation; Behavioral: Usual care genetics referral
- Usual care breast cancer screening navigation + pretest education/usual care genetic referral (Experimental)
  Interventions: Behavioral: Breast cancer screening navigation; Behavioral: Pretest education + usual care genetics referral
- Multicancer screening navigation + usual care genetic referral (Experimental)
  Interventions: Behavioral: Multicancer screening navigation; Behavioral: Usual care genetics referral
- Multicancer screening navigation + pretest education/usual care genetic referral (Experimental)
  Interventions: Behavioral: Multicancer screening navigation; Behavioral: Pretest education + usual care genetics referral

INTERVENTIONS:
Behavioral: Breast cancer screening navigation — Single cancer navigation includes the following, oriented to breast cancer only: cancer education, barrier assessment and resolution, screening exam scheduling, text and mail reminders, documentation of appointment completion and results communicated to patient.
  Arms: Usual care breast cancer screening navigation; Usual care breast cancer screening navigation + pretest education/usual care genetic referral; Usual care breast cancer screening navigation + usual care genetic referral
Behavioral: Multicancer screening navigation — Multi-cancer navigation includes the following, oriented to breast and colorectal cancers: cancer education, barrier assessment and resolution, screening exam scheduling, text and mail reminders, documentation of appointment completion and results communicated to patient.
  Arms: Multicancer screening navigation; Multicancer screening navigation + pretest education/usual care genetic referral; Multicancer screening navigation + usual care genetic referral
Behavioral: Usual care genetics referral — Referral for genetics will be provided at the completion of the navigation call.
  Arms: Multicancer screening navigation + usual care genetic referral; Usual care breast cancer screening navigation + usual care genetic referral
Behavioral: Pretest education + usual care genetics referral — Print education regarding the genetic counseling and testing process and specific tips to support at-home testing. Referral for genetics will be provided at the completion of the navigation call.
  Arms: Multicancer screening navigation + pretest education/usual care genetic referral; Usual care breast cancer screening navigation + pretest education/usual care genetic referral

SUMMARY:
The goal of this study is to test bundled familial cancer risk assessment + multicancer (colorectal + breast) vs. single (breast) cancer navigation, using a wait list control for colorectal cancer screening referral and navigation. Among those eligible, this study will test usual care referral to genetic services vs. pretest education + usual care referral. The study also will assess how bundled multicancer navigation works and for whom it is most effective through a multisite, mixed-methods patient- and organization-level process evaluation.

DETAILED DESCRIPTION:
Research Design and Methods:

All women referred for screening navigation within community navigation programs receive familial cancer risk assessment, bundled with either multicancer (colorectal + breast) vs. single (breast) cancer navigation, with a wait list control for colorectal cancer screening referral and navigation, stratified by site and genetics referral eligibility. Primary analyses will be conducted among those randomized to multicancer or single cancer navigation, but ineligible for genetic referral, to test effectiveness for colorectal cancer screening and non-inferiority for breast cancer screening (N=600). In exploratory subanalyses among those referred to genetic counseling based on their familial cancer risk assessment, the study will test the effect of four bundles that combine multicancer vs. single cancer navigation with usual care referral to telephone-based pretest and posttest genetic counseling and testing or video and print pre-counseling education + referral (N=180). A multi-site, mixed-methods organization- and patient-focused process evaluation is conducted alongside and at the conclusion of the trial.

Research Procedures:

Research staff not associated with navigation programs will obtain consent and HIPAA authorization, proceeding with baseline assessment and randomization, stratified by site and genetics eligibility. The trial will recruit (N=820) and retain (N=780) women to this trial within two years. N=600 are retained for primary analyses; N=180 are retained for exploratory outcomes among those referred to genetic services.

Randomization. At the end of the baseline assessment, research staff randomize participants to the single or multicancer navigation conditions, stratified by navigation site and genetic testing eligibility. Participants will be notified of study condition and connected to a navigator. Participants eligible for genetic services will receive services related to their study arm from their navigator following completion of multicancer or single cancer screening navigation. This will result in four bundles of screening and genetic services to be assessed in exploratory analyses. Contamination is mitigated through navigator training and supervision and documentation tracking. Participants will be randomized in blocks of 4 or 6 to support equal sample sizes across arms.

Navigation Protocol. Guided stepwise protocols ensure documentation and timeliness of navigation and address contamination during navigation. Steps are chronological; navigators document completion of a step to move to the next. Wait-list navigation for those in the single cancer navigation arm who have not received colorectal cancer screening by 6-months will receive colorectal cancer screening referral and navigation at this time.

ELIGIBILITY:
Inclusion Criteria:

1. Seeking screening navigation services through programs at a participating site (Georgetown Lombardi Cancer Center or Helen F. Graham Cancer Center & Research Institutes)
2. Eligible for breast cancer screening while also due and eligible for colorectal cancer screening (per USPSTF guidelines)
3. Female sex
4. Aged 45-74
5. Identify as Black/African American race and/or Hispanic/Latin(e)(a) ethnicity
6. Speak English or Spanish with enough fluency to complete study activities
7. Stated willingness to comply with all study procedures (navigation, surveys) and availability for the duration of the study
8. Provision of completed electronic informed consent form

Exclusion Criteria:

1. Not engaged with or planning to use navigation programs at Georgetown Lombardi Cancer Center and Helen F. Graham Cancer Center & Research Institute
2. Not eligible for breast cancer screening or not due and eligible for colorectal cancer screening (per USPSTF guidelines)
3. History of breast and/or colorectal cancer; or Reporting symptoms related to breast and/or colorectal cancer (e.g., GI bleeding, breast mass)
4. Male sex, Intersex, or other sex
5. Under age 45 or over age 74
6. Identifies as neither Black/African American race nor Hispanic/Latin(e)(a) ethnicity
7. Speaks neither English nor Spanish with enough fluency to complete study activities
8. Stated unwillingness to comply with study procedures (navigation, surveys) or unavailability for the duration of the study
9. Inability to provide electronic informed consent, or needing another person to authorize informed consent on their behalf

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Receipt of colorectal cancer screening | 6 months after navigation completion
  Colorectal cancer screening will be determined through electronic health records abstraction. Documentation of screening includes the test (FIT, colonoscopy), date, clinical indication, assessment or result (imaging, pathology) and recommendations and procedures as applicable, following to treatment initiation.
Receipt of breast cancer screening | Six months after completion of navigation
  Breast cancer screening (mammography, tomosynthesis, MRI, breast ultrasound, breast biopsy) will be determined through electronic health records abstraction. Documentation of screening includes the test, date, clinical indication, assessment or result (imaging, pathology) and recommendations and procedures as applicable, following to treatment initiation.

OTHER OUTCOMES:
Receipt of genetic testing | Six months after completion of navigation
  Receipt of genetic testing as well as posttest genetic counseling within 6 months of randomization; documentation of test, test result, date, will be drawn from electronic health records
Receipt of genetic counseling | Six months after completion of navigation
  Documented attendance/date of pretest genetic counseling appointment within 6 months of randomization

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - ChristianaCare-Helen F. Graham Cancer Center & Research Institute, Newark, Delaware
  - Georgetown University, Washington D.C., District of Columbia